CLINICAL TRIAL: NCT04929483
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Tolerability of BIO89-100 in Subjects With Biopsy-Confirmed Nonalcoholic Steatohepatitis (NASH)
Brief Title: Study Evaluating the Safety, Efficacy and Tolerability of BIO89-100 in Subjects With Biopsy-confirmed Nonalcoholic Steatohepatitis (NASH)
Acronym: ENLIVEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 89bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO89-100-122
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: Liver Diseases; Fatty Liver; Digestive System Diseases; Non-alcoholic Fatty Liver Disease; Metabolic diseases; MASH MAFLD; NASH NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fatty Liver; Digestive System Diseases; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- BIO89-100 - 15 mg once weekly (QW) (Experimental)
  Interventions: Drug: BIO89-100
- BIO89-100 - 30 mg QW (Experimental)
  Interventions: Drug: BIO89-100
- BIO89-100 - 44 mg once every 2 weeks (Q2W) (Experimental)
  Interventions: Drug: BIO89-100
- Placebo QW (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo Q2W (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo QW (Main study)/ BIO89-100 - 30 mg QW (Extension) (Experimental)
  Interventions: Drug: BIO89-100; Drug: Placebo

INTERVENTIONS:
Drug: BIO89-100 — Subcutaneous injection
  Other Names: Pegozafermin
  Arms: BIO89-100 - 15 mg once weekly (QW); BIO89-100 - 30 mg QW; BIO89-100 - 44 mg once every 2 weeks (Q2W); Placebo QW (Main study)/ BIO89-100 - 30 mg QW (Extension)
Drug: Placebo — Subcutaneous injection
  Arms: Placebo Q2W; Placebo QW; Placebo QW (Main study)/ BIO89-100 - 30 mg QW (Extension)

SUMMARY:
This is a randomized, double-blind, placebo-controlled study that will evaluate the safety, efficacy, tolerability of BIO89-100 in patients with biopsy-confirmed fibrosis stages F2-F3 NASH.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 21 to 75
* Biopsy-confirmed NASH with fibrosis stage F2 or F3 per NASH CRN System and NAS ≥4, with a score of at least 1 in each of steatosis, ballooning degeneration, and lobular inflammation.

  * Qualifying biopsy must be either within 6 months of screening visit or obtained during screening period

Key Exclusion Criteria:

* Have poorly controlled high blood pressure
* Have type 1 diabetes or poorly controlled type 2 diabetes.
* History of cirrhosis or evidence of cirrhosis by clinical, imaging, or liver biopsy evaluation
* Are planning to try to lose weight during the conduct of the study.
* Have a BMI <25 kg/m2

Other inclusion and exclusion criteria may apply.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Millie Gottwald, PharmD, Study Director — 89bio, Inc.
Locations (72):
- United States (71):
  - 89bio Clinical Study Site, Birmingham, Alabama
  - 89bio Clinical Study Site, Dothan, Alabama
  - 89bio Clinical Study Site, Guntersville, Alabama
  - 89bio Clinical Study Site, Madison, Alabama
  - 89bio Clinical Study Site, Chandler, Arizona
  - 89bio Clinical Study Site, Glendale, Arizona
  - 89bio Clinical Study Site, Peoria, Arizona
  - 89bio Clinical Study Site, Tucson, Arizona
  - 89bio Clinical Study Site, Little Rock, Arkansas
  - 89bio Clinical Study Site, Chula Vista, California
  - 89bio Clinical Study Site, Huntington Park, California
  - 89bio Clinical Study Site, Long Beach, California
  - 89bio Clinical Study Site, Orange, California
  - 89bio Clinical Study Site, Panorama City, California
  - 89bio Clinical Study Site, Rialto, California
  - 89bio Clinical Study Site, Santa Ana, California
  - 89bio Clinical Study Site, Englewood, Colorado
  - 89bio Clinical Study Site, Boynton Beach, Florida
  - 89bio Clinical Study Site, Bradenton, Florida
  - 89bio Clinical Study Site, Fort Myers, Florida
  - 89bio Clinical Study Site, Lakeland, Florida
  - 89bio Clinical Study Site, Maitland, Florida
  - 89bio Clinical Study Site, Miami, Florida
  - 89bio Clinical Study Site, Miami Lakes, Florida
  - 89bio Clinical Study Site, Ocala, Florida
  - 89bio Clinical Study Site, Palmetto Bay, Florida
  - 89bio Clinical Study Site, Pinellas Park, Florida
  - 89bio Clinical Study Site, Port Orange, Florida
  - 89bio Clinical Study Site, Sarasota, Florida
  - 89bio Clinical Study Site, Viera, Florida
  - 89bio Clinical Study Site, Athens, Georgia
  - 89bio Clinical Study Site, Sandy Springs, Georgia
  - 89bio Clinical Study Site, New Albany, Indiana
  - 89bio Clinical Study Site, South Bend, Indiana
  - 89bio Clinical Study Site, Iowa City, Iowa
  - 89bio Clinical Study Site, Topeka, Kansas
  - 89bio Clinical Study Site, Marrero, Louisiana
  - 89bio Clinical Study Site, Monroe, Louisiana
  - 89bio Clinical Study Site, Shreveport, Louisiana
  - 89bio Clinical Study Site, Glen Burnie, Maryland
  - 89bio Clinical Study Site, Greenbelt, Maryland
  - 89bio Clinical Study Site, St Louis, Missouri
  - 89bio Clinical Study Site, Las Vegas, Nevada
  - 89bio Clinical Study Site, Florham Park, New Jersey
  - 89bio Clinical Study Site, New York, New York
  - 89bio Clinical Study Site, Concord, North Carolina
  - 89bio Clinical Study Site, Columbus, Ohio
  - 89bio Clinical Study Site, Dayton, Ohio
  - 89bio Clinical Study Site, Springboro, Ohio
  - 89bio Clinical Study Site, Westlake, Ohio
  - 89bio Clinical Study Site, Greenwood, South Carolina
  - 89bio Clinical Study Site, Summerville, South Carolina
  - 89bio Clinical Study Site, Chattanooga, Tennessee
  - 89bio Clinical Study Site, Hermitage, Tennessee
  - 89bio Clinical Study Site, Austin, Texas
  - 89bio Clinical Study Site, Beaumont, Texas
  - 89bio Clinical Study Site, Dallas, Texas
  - 89bio Clinical Study Site, Edinburg, Texas
  - 89bio Clinical Study Site, Fort Worth, Texas
  - 89bio Clinical Study Site, Garland, Texas
  - 89bio Clinical Study Site, Houston, Texas
  - 89bio Clinical Study Site, San Antonio, Texas
  - 89bio Clinical Study Site, Waco, Texas
  - 89bio Clinical Study Site, Wichita Falls, Texas
  - 89bio Clinical Study Site, Ogden, Utah
  - 89bio Clinical Study Site, Sandy City, Utah
  - 89bio Clinical Study Site, Manassas, Virginia
  - 89bio Clinical Study Site, Richmond, Virginia
  - 89bio Clinical Study Site, Roanoke, Virginia
  - 89bio Clinical Study Site, Seattle, Washington
  - 89bio Clinical Study Site, Spokane, Washington
- 89bio Clinical Study Site, San Juan, Puerto Rico

REFERENCES:
- [Derived] Tseng CL, Balic K, Charlton RW, Margalit M, Mansbach H, Savic RM. Population Pharmacokinetics and Pharmacodynamics of Pegozafermin in Patients with Nonalcoholic Steatohepatitis. Clin Pharmacol Ther. 2023 Dec;114(6):1323-1331. doi: 10.1002/cpt.3046. Epub 2023 Oct 2. PMID 37696614
- [Derived] Loomba R, Sanyal AJ, Kowdley KV, Bhatt DL, Alkhouri N, Frias JP, Bedossa P, Harrison SA, Lazas D, Barish R, Gottwald MD, Feng S, Agollah GD, Hartsfield CL, Mansbach H, Margalit M, Abdelmalek MF. Randomized, Controlled Trial of the FGF21 Analogue Pegozafermin in NASH. N Engl J Med. 2023 Sep 14;389(11):998-1008. doi: 10.1056/NEJMoa2304286. Epub 2023 Jun 24. PMID 37356033

RESULTS

PARTICIPANT FLOW:
Groups:
- Main and Extension Study: Pegozafermin 15 mg QW: Participants received pegozafermin 15 milligrams (mg) once weekly (QW) as a subcutaneous (SC) injection for 24 weeks in the main study and for 24 weeks in the extension study.
- Main and Extension Study: Pegozafermin 30 mg QW: Participants received pegozafermin 30 mg QW as a SC injection for 24 weeks in the main study and for 24 weeks in the extension study.
- Main and Extension Study: Pegozafermin 44 mg Q2W: Participants received pegozafermin 44 mg every 2 weeks (Q2W) as a SC injection for 24 weeks in the main study and for 24 weeks in the extension study.
- Main Study: Placebo Pooled: Participants received placebo matched to pegozafermin QW or Q2W as a SC injection for 24 weeks in the main study.
- Main and Extension Study: Placebo (Main) and Placebo (Extension) Only: Participants who received placebo QW as a SC injection for 24 weeks in the main study were re-randomized to receive placebo QW as a SC injection for 24 weeks in the extension study. Participants who received placebo Q2W as a SC injection for 24 weeks in the main study continued on placebo Q2W for 24 weeks in the extension study.
- Main and Extension Study: Placebo (Main) and Pegozafermin 30 mg QW (Extension): Participants who received placebo QW in the main study were re-randomized to receive pegozafermin 30 mg QW as a SC injection for 24 weeks in the extension study.
Period: Main Study (24 Weeks)
Arm/Group | Main and Extension Study: Pegozafermin 15 mg QW | Main and Extension Study: Pegozafermin 30 mg QW | Main and Extension Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled | Main and Extension Study: Placebo (Main) and Placebo (Extension) Only | Main and Extension Study: Placebo (Main) and Pegozafermin 30 mg QW (Extension)
Started | 21 | 73 | 57 | 71 | 0 | 0
Received at Least 1 Dose of Study Drug | 21 | 72 | 57 | 69 | 0 | 0
Safety Analysis Set | 21 | 72 | 57 | 69 | 0 | 0
Pharmacokinetic (PK) Analysis Set | 14 | 66 | 51 | 0 | 0 | 0
MRI-PDFF Analysis Set | 14 | 61 | 49 | 57 | 0 | 0
Full Analysis Set | 14 | 66 | 51 | 61 | 0 | 0
Completed | 20 | 59 | 51 | 63 | 0 | 0
Not Completed | 1 | 14 | 6 | 8 | 0 | 0
Not completed — Adverse Event | 1 | 6 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 3 | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Randomized in error | 0 | 1 | 0 | 2 | 0 | 0
Period: Extension Study (24 Weeks)
Arm/Group | Main and Extension Study: Pegozafermin 15 mg QW | Main and Extension Study: Pegozafermin 30 mg QW | Main and Extension Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled | Main and Extension Study: Placebo (Main) and Placebo (Extension) Only | Main and Extension Study: Placebo (Main) and Pegozafermin 30 mg QW (Extension)
Started | 20 | 56 | 50 | 0 | 42 | 19
Received at Least 1 Dose of Study Drug | 20 | 56 | 48 | 0 | 42 | 19
Completed | 19 | 53 | 42 | 0 | 38 | 19
Not Completed | 1 | 3 | 8 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Other than specified | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized analysis set included all enrolled participants who were assigned a randomization number in the study.
Groups:
- Main and Extension Study: Pegozafermin 15 mg QW: Participants received pegozafermin 15 mg QW as a SC injection for 24 weeks in the main study and for 24 weeks in the extension study.
- Main and Extension Study: Pegozafermin 44 mg Q2W: Participants received pegozafermin 44 mg Q2W as a SC injection for 24 weeks in the main study and for 24 weeks in the extension study.
- Total: Total of all reporting groups
Arm/Group | Main and Extension Study: Pegozafermin 15 mg QW | Main and Extension Study: Pegozafermin 30 mg QW | Main and Extension Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled | Total
Number analyzed (Participants) | 21 | 73 | 57 | 71 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (10.45) | 55.3 (11.15) | 55.2 (11.23) | 56.3 (9.01) | 55.6 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 50 | 20 | 39 | 118
  Male | 12 | 23 | 37 | 32 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 32 | 20 | 24 | 85
  Not Hispanic or Latino | 12 | 41 | 37 | 47 | 137
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 3 | 0 | 0 | 4
  White | 18 | 69 | 54 | 67 | 208
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Number of Participants With Histological Resolution of Nonalcoholic Steatohepatitis (NASH) Without Worsening of Fibrosis
Description: Nonalcoholic fatty liver disease activity score (NAS) was the sum of the scores of steatosis, inflammation, and ballooning. NAS score ranged from 0 to 8, with higher scores indicating worse disease severity. Resolution of NASH was defined as the total absence of ballooning (score=0) and absent or mild inflammation (score=0 to 1). NASH clinical research system (CRN) fibrosis is staged on a 0-4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis). Worsening of fibrosis was defined as progression of fibrosis greater than or equal to (≥) 1 stage in NASH CRN fibrosis score.
Time Frame: Week 24
Population: Full analysis set (FAS) included all enrolled participants with confirmed fibrosis stage F2 or F3 and NAS ≥4 at baseline per independent review by a 3-pathologist panel who were eligible and assigned a randomization number in the study and received at least 1 dose of investigational product (IP). Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Main Study: Pegozafermin 15 mg QW: Participants received pegozafermin 15 mg QW as a SC injection for 24 weeks.
- Main Study: Pegozafermin 30 mg QW: Participants received pegozafermin 30 mg QW as a SC injection for 24 weeks.
- Main Study: Pegozafermin 44 mg Q2W: Participants received pegozafermin 44 mg Q2W as a SC injection for 24 weeks.
- Main Study: Placebo Pooled: Participants received placebo matched to pegozafermin QW or Q2W as a SC injection for 24 weeks.
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled
Number analyzed (Participants) | 14 | 53 | 43 | 54
Participants | 5 | 12 | 11 | 1
Statistical Analysis 1: Comparison: Main Study: Pegozafermin 15 mg QW vs Main Study: Placebo Pooled; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel with missing outcome measures handled by multiple imputation method; Treatment Difference = 34.65, 95% CI 2-sided [10.04 to 59.26]
Statistical Analysis 2: Comparison: Main Study: Pegozafermin 30 mg QW vs Main Study: Placebo Pooled; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel with missing outcome measures handled by multiple imputation method; Treatment Difference = 20.89, 95% CI 2-sided [9.05 to 32.72]
Statistical Analysis 3: Comparison: Main Study: Pegozafermin 44 mg Q2W vs Main Study: Placebo Pooled; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel with missing outcome measures handled by multiple imputation method; Treatment Difference = 23.61, 95% CI 2-sided [10.04 to 37.18]

2. Primary Outcome: Main Study: Number of Participants Who Achieved Improvement of Fibrosis ≥1 Stage Without Worsening of NASH
Description: Worsening of NASH was defined as increase in nonalcoholic fatty liver disease activity score (NAS) for ballooning, inflammation, or steatosis. NAS was the sum of the scores of steatosis, inflammation, and ballooning. NAS score ranged from 0 to 8, with higher scores indicating worse disease severity. Fibrosis improvement was defined as ≥1-stage decrease in NASH CRN fibrosis score. NASH CRN fibrosis was staged on a 0-4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis).
Time Frame: Week 24
Population: FAS included all enrolled participants with confirmed fibrosis stage F2 or F3 and NAS ≥4 at baseline per independent review by a 3-pathologist panel who were eligible and assigned a randomization number in the study and received at least 1 dose of IP. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled
Number analyzed (Participants) | 14 | 53 | 43 | 54
Participants | 3 | 14 | 11 | 4
Statistical Analysis 1: Comparison: Main Study: Pegozafermin 15 mg QW vs Main Study: Placebo Pooled; Test type: Superiority; p = 0.1039, Cochran-Mantel-Haenszel; Treatment Difference = 14.45, 95% CI 2-sided [-8.71 to 37.62]
Statistical Analysis 2: Comparison: Main Study: Pegozafermin 30 mg QW vs Main Study: Placebo Pooled; Test type: Superiority; p = 0.0085, Cochran-Mantel-Haenszel; Treatment Difference = 18.87, 95% CI 2-sided [5.24 to 32.50]
Statistical Analysis 3: Comparison: Main Study: Pegozafermin 44 mg Q2W vs Main Study: Placebo Pooled; Test type: Superiority; p = 0.0077, Cochran-Mantel-Haenszel; Treatment Difference = 20.33, 95% CI 2-sided [5.26 to 35.40]

3. Secondary Outcome: Main Study: Number of Participants With at Least a 2-Point Improvement in NAS and no Worsening of Fibrosis
Description: NAS was the sum of the scores of steatosis, inflammation, and ballooning. NAS score ranged from 0 to 8, with higher scores indicating worse disease severity. Worsening of fibrosis was defined as progression of fibrosis ≥1 stage in NASH CRN fibrosis score. NASH CRN fibrosis is staged on a 0-4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis).
Time Frame: Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled
Number analyzed (Participants) | 14 | 53 | 43 | 54
Participants | 5 | 34 | 26 | 13

4. Secondary Outcome: Main Study: Number of Participants With NASH Resolution and Fibrosis Improvement ≥1 Stage
Description: NAS was the sum of the scores of steatosis, inflammation, and ballooning. NAS score ranged from 0 to 8, with higher scores indicating worse disease severity. Resolution of NASH was defined as the total absence of ballooning (score=0) and absent or mild inflammation (score=0 to 1). Fibrosis improvement was defined as ≥1-stage decrease in NASH CRN fibrosis score. NASH CRN fibrosis was staged on a 0-4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis).
Time Frame: Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled
Number analyzed (Participants) | 14 | 53 | 43 | 54
Participants | 2 | 7 | 8 | 0

5. Secondary Outcome: Main Study: Number of Participants With at Least a 2-point Improvement in NAS Score and Are Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF) Responders and Alanine Aminotransferase (ALT) Responders
Description: A responder was defined as achieving ≥2 point improvement in NAS score and are MRI-PDFF responders and ALT responders at Week 24. NAS was the sum of the scores of steatosis, inflammation, and ballooning. NAS score ranged from 0 to 8, with higher scores indicating worse disease severity. MRI-PDFF responder was defined as ≥30% reduction from baseline in liver fat by MRI-PDFF. ALT responder was defined as ≥17 units/liter (U/L) or ≥30% reduction from baseline in ALT.
Time Frame: Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled
Number analyzed (Participants) | 14 | 53 | 43 | 54
Participants | 4 | 31 | 22 | 5

6. Secondary Outcome: Main Study: Percent Change From Baseline in Serum Triglycerides
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled
Number analyzed (Participants) | 12 | 57 | 45 | 57
Percent change | -5.79 (19.473) | -14.87 (54.765) | -7.79 (29.612) | 1.02 (31.425)

7. Secondary Outcome: Main Study: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-c)
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled
Number analyzed (Participants) | 11 | 55 | 44 | 56
Percent change | 20.28 (74.840) | -0.42 (35.290) | -5.64 (31.944) | 0.32 (30.811)

8. Secondary Outcome: Main Study: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-c)
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled
Number analyzed (Participants) | 12 | 57 | 45 | 57
Percent change | -3.04 (18.421) | -6.94 (21.260) | -6.95 (24.120) | -0.46 (24.081)

9. Secondary Outcome: Main Study: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-c)
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled
Number analyzed (Participants) | 12 | 57 | 45 | 57
Percent change | 4.69 (13.441) | 15.82 (20.376) | 7.31 (18.690) | -2.01 (13.592)

10. Secondary Outcome: Main Study: Percent Change From Baseline in Adiponectin
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled
Number analyzed (Participants) | 13 | 56 | 46 | 57
Percent change | 22.73 (44.045) | 31.36 (49.215) | 26.60 (46.353) | -6.28 (23.770)

11. Secondary Outcome: Main Study: Percent Change From Baseline in HbA1c (Glycated Hemoglobin)
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Pooled
Number analyzed (Participants) | 14 | 57 | 45 | 56
Percent change | -2.24 (13.039) | -3.74 (11.216) | -2.00 (11.742) | -0.52 (9.012)

12. Secondary Outcome: Main Study: Percent Change From Baseline in Alanine Transaminase
Time Frame: Baseline, Week 12 and 24
Population: FAS included all enrolled participants with confirmed fibrosis stage F2 or F3 and NAS ≥4 at baseline per independent review by a 3-pathologist panel who were eligible and assigned a randomization number in the study and received at least 1 dose of IP. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable for specified time points.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Main Study: Placebo Only Pooled: Participants received placebo matched to pegozafermin QW or Q2W as a SC injection for 24 weeks.
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Only Pooled
Number analyzed (Participants) | 14 | 61 | 47 | 57
Percent change
  Change at Week 12 | -39.68 (33.615) | -42.04 (23.044) | -35.42 (28.874) | -8.62 (35.051)
  Change at Week 24: number analyzed (Participants) | 13 | 57 | 46 | 57
  Change at Week 24 | -39.28 (31.478) | -42.73 (25.218) | -31.33 (43.053) | -0.41 (48.798)

13. Secondary Outcome: Main Study: Percent Change From Baseline in Hepatic Fat Fraction By Magnetic Resonance Imaging - (MRI-PDFF)
Time Frame: Baseline, Week 12 and 24
Population: MRI-PDFF analysis set included all participants in the FAS who had a baseline and at least one follow-up MRI-PDFF assessment. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable for specified time points.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Main Study: Placebo Only Pooled: Participants who received placebo QW or Q2W as a SC injection for 24 weeks.
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Only Pooled
Number analyzed (Participants) | 14 | 61 | 49 | 57
Percent Change
  Change at Week 12: number analyzed (Participants) | 14 | 61 | 49 | 53
  Change at Week 12 | -45.05 (25.857) | -57.07 (19.563) | -50.63 (21.225) | -0.53 (42.062)
  Change at Week 24: number analyzed (Participants) | 14 | 54 | 45 | 57
  Change at Week 24 | -27.92 (35.209) | -51.05 (24.065) | -42.90 (40.257) | -5.80 (47.605)

14. Secondary Outcome: Main Study: Percent Change From Baseline in N-Terminal Type III Collagen Propeptide (Pro-C3)
Time Frame: Baseline, Week 12 and 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W | Main Study: Placebo Only Pooled
Number analyzed (Participants) | 13 | 62 | 49 | 55
Percent Change
  Change at Week 12 | -35.34 (26.673) | -9.51 (37.151) | -13.84 (25.420) | 10.57 (33.392)
  Change at Week 24: number analyzed (Participants) | 13 | 56 | 45 | 55
  Change at Week 24 | -17.10 (34.345) | -17.76 (28.250) | -15.22 (27.429) | 9.46 (45.403)

15. Secondary Outcome: Main Study: Trough Serum Concentration of Pegozafermin
Description: Serum trough concentration (ng/mL) of pegozafermin taken from pre-dose samples.
Time Frame: Predose at Week 12 and 24
Population: Pharmacokinetic analysis set included all participants in the FAS who had sufficient data to adequately characterize the trough serum pegozafermin concentrations and had no other events or protocol violations that would adversely affect results, such as not completing the full dose. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable for specified time points.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | Main Study: Pegozafermin 15 mg QW | Main Study: Pegozafermin 30 mg QW | Main Study: Pegozafermin 44 mg Q2W
Number analyzed (Participants) | 13 | 50 | 36
nanograms/milliliter
  Week 12: number analyzed (Participants) | 11 | 50 | 36
  Week 12 | 197.833 (110.097) | 534.289 (375.149) | 81.699 (77.099)
  Week 24: number analyzed (Participants) | 13 | 38 | 30
  Week 24 | 168.127 (158.749) | 691.424 (718.495) | 84.033 (77.896)

16. Secondary Outcome: Main and Extension Study: Percent Change From Baseline in Alanine Transaminase
Description: Baseline was prior to dosing on Day 1 of the main study.
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Main and Extension Study: Pegozafermin 15 mg QW | Main and Extension Study: Pegozafermin 30 mg QW | Main and Extension Study: Pegozafermin 44 mg Q2W | Main and Extension Study: Placebo (Main) and Placebo (Extension) Only | Main and Extension Study: Placebo (Main) and Pegozafermin 30 mg QW (Extension)
Number analyzed (Participants) | 14 | 48 | 38 | 32 | 19
Percent change | -28.51 (37.164) | -45.08 (25.068) | -38.05 (28.256) | -5.03 (43.918) | -31.71 (46.868)

17. Secondary Outcome: Main and Extension Study: Percent Change From Baseline in N-Terminal Type III Collagen Propeptide (Pro-C3)
Description: Baseline was prior to dosing on Day 1 of the main study.
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Main and Extension Study: Pegozafermin 15 mg QW | Main and Extension Study: Pegozafermin 30 mg QW | Main and Extension Study: Pegozafermin 44 mg Q2W | Main and Extension Study: Placebo (Main) and Placebo (Extension) Only | Main and Extension Study: Placebo (Main) and Pegozafermin 30 mg QW (Extension)
Number analyzed (Participants) | 13 | 47 | 37 | 32 | 18
Percent Change | -7.89 (21.069) | -16.82 (23.675) | -14.96 (21.342) | 1.64 (33.082) | -17.22 (23.053)

18. Secondary Outcome: Main and Extension Study: Percent Change From Baseline in Hepatic Fat Fraction By Magnetic Resonance Imaging - (MRI-PDFF)
Description: Baseline was prior to dosing on Day 1 of the main study.
Time Frame: Baseline, Week 48
Population: MRI-PDFF analysis set included all participants in the FAS who had a baseline and at least one follow-up MRI-PDFF assessment. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Main and Extension Study: Pegozafermin 15 mg QW | Main and Extension Study: Pegozafermin 30 mg QW | Main and Extension Study: Pegozafermin 44 mg Q2W | Main and Extension Study: Placebo (Main) and Placebo (Extension) Only | Main and Extension Study: Placebo (Main) and Pegozafermin 30 mg QW (Extension)
Number analyzed (Participants) | 13 | 48 | 40 | 32 | 19
Percent Change | -23.93 (33.557) | -48.75 (29.717) | -25.93 (50.980) | -3.15 (47.992) | -59.14 (25.807)

19. Secondary Outcome: Main and Extension Study: Trough Serum Concentration of Pegozafermin
Description: Serum trough concentration (ng/mL) of pegozafermin taken from pre-dose samples.
Time Frame: Predose at Week 48
Population: Pharmacokinetic analysis set included all participants in the FAS who had sufficient data to adequately characterize the trough serum pegozafermin concentrations and had no other events or protocol violations that would adversely affect results, such as not completing the full dose. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | Main and Extension Study: Pegozafermin 15 mg QW | Main and Extension Study: Pegozafermin 30 mg QW | Main and Extension Study: Pegozafermin 44 mg Q2W | Main and Extension Study: Placebo (Main) and Pegozafermin 30 mg QW (Extension)
Number analyzed (Participants) | 10 | 35 | 25 | 10
nanograms/milliliter | 206.54 (93.104) | 471.28 (397.691) | 111.00 (88.644) | 553.45 (651.882)

20. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of IP, whether or not considered related to the IP. TEAEs were defined as AEs that started or worsened on or after the first dose of study IP up to Week 51. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect, important medical event or reaction. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Week 51
Population: Safety analysis set included all randomized participants who received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Main and Extension Study: Pegozafermin 15 mg QW | Main and Extension Study: Pegozafermin 30 mg QW | Main and Extension Study: Pegozafermin 44 mg Q2W | Main and Extension Study: Placebo (Main) and Placebo (Extension) Only | Main and Extension Study: Placebo (Main) and Pegozafermin 30 mg QW (Extension)
Number analyzed (Participants) | 21 | 72 | 57 | 50 | 19
Participants
  TEAEs | 21 | 63 | 46 | 42 | 17
  SAEs | 1 | 5 | 8 | 6 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to Week 51
Description: Safety analysis set included all randomized participants who received at least 1 dose of IP. As pre-specified, data for the placebo arm was combined for the main and extension study.
Arm/Group | Main and Extension Study: Pegozafermin 15 mg QW | Main and Extension Study: Pegozafermin 30 mg QW | Main and Extension Study: Pegozafermin 44 mg Q2W | Main and Extension Study: Placebo (Main) and Placebo (Extension) Only | Main and Extension Study: Placebo (Main) and Pegozafermin 30 mg QW (Extension)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/72 | 0/57 | 0/50 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/21 | 5/72 | 8/57 | 6/50 | 2/19
Other Adverse Events (participants affected / at risk) | 21/21 | 62/72 | 45/57 | 41/50 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main and Extension Study: Pegozafermin 15 mg QW (N=21) | Main and Extension Study: Pegozafermin 30 mg QW (N=72) | Main and Extension Study: Pegozafermin 44 mg Q2W (N=57) | Main and Extension Study: Placebo (Main) and Placebo (Extension) Only (N=50) | Main and Extension Study: Placebo (Main) and Pegozafermin 30 mg QW (Extension) (N=19)
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Brain stem haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Spinal claudication (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main and Extension Study: Pegozafermin 15 mg QW (N=21) | Main and Extension Study: Pegozafermin 30 mg QW (N=72) | Main and Extension Study: Pegozafermin 44 mg Q2W (N=57) | Main and Extension Study: Placebo (Main) and Placebo (Extension) Only (N=50) | Main and Extension Study: Placebo (Main) and Pegozafermin 30 mg QW (Extension) (N=19)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 5 | 1 | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 8 | 3 | 4 | 2
Abdominal pain lower (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 3 | 5 | 1
Constipation (Gastrointestinal disorders) | 0 | 5 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 18 | 9 | 5 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 5 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 26 | 11 | 5 | 5
Vomiting (Gastrointestinal disorders) | 2 | 13 | 2 | 2 | 2
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 1 | 4 | 3 | 5 | 2
Injection site erythema (General disorders) | 3 | 11 | 3 | 3 | 2
Injection site pain (General disorders) | 0 | 1 | 1 | 1 | 1
Injection site pruritus (General disorders) | 0 | 6 | 3 | 0 | 4
Injection site rash (General disorders) | 0 | 7 | 2 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 0 | 2 | 2
Vaccination site joint pain (General disorders) | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 4 | 14 | 8 | 9 | 3
Ear infection (Infections and infestations) | 0 | 0 | 3 | 2 | 0
Influenza (Infections and infestations) | 1 | 0 | 2 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 4 | 8 | 2 | 2
Tooth infection (Infections and infestations) | 2 | 2 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 10 | 2 | 4 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 1
Procedural pain (Injury, poisoning and procedural complications) | 4 | 0 | 1 | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cortisol increased (Investigations) | 0 | 0 | 0 | 3 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 5 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Increased appetite (Metabolism and nutrition disorders) | 2 | 11 | 4 | 2 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 7 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 2 | 1
Headache (Nervous system disorders) | 2 | 6 | 6 | 3 | 4
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 2 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 4 | 2 | 2 | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT04929483/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT04929483/SAP_001.pdf